CLINICAL TRIAL: NCT02949245
Title: Evaluation of Neurologic Complications Associated With Surgical Correction of Adult Spinal Deformity (Scoli-RISK-1): A Prospective, Observational, Multi-center Study 5 Year Follow-up Extension
Brief Title: Neurologic Complications in Spinal Deformity Surgery - Extension
Status: Completed | Type: Observational
Sponsor: AO Foundation, AO Spine (Other)
Collaborators: Scoliosis Research Society (Other)
Responsible Party: Sponsor
Other Study IDs: Scoli-RISK-1 extension
Record Dates: First submitted 2016-10-24; First posted 2016-10-31 (Estimated); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Adult Spinal Deformity
Keywords: Spine; Surgery; Prospective Studies; Deformity; Neurologic deficit
MeSH Terms: conditions — Congenital Abnormalities; Neurologic Manifestations | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Groups/Cohorts: Surgical treatment
  This observational study is examining the outcomes of standard surgical treatments for adult spinal deformity.
  Interventions: Procedure: Interventions

INTERVENTIONS:
Procedure: Interventions — Procedure/Surgery: Routinely performed surgical correction of spinal deformity
  Routinely performed surgical correction of spinal deformity

SUMMARY:
272 subjects with "high risk" adult spinal deformity requiring surgical correction were enrolled in the previous prospective multi-center international Scoli-RISK-1 study. "High risk" patients were defined by either their diagnoses and/or the type of surgical intervention as listed in the inclusion criteria. Neurological complications in the form of new motor and sensory deficits were monitored prospectively in all patients at hospital discharge, at 6 weeks (± 2 weeks), 6 months (± 2 months) and 24 months (± 2 months) after the surgery. The relationship to the surgical intervention was assessed in all new deficits.

Regression analyses were used to evaluate the association between patient demographics, co-morbidities, treatment history, spinal deformity characteristics, surgical characteristics, non-neurologic complications and pre-surgical status to occurrence of a neurologic deficit after surgery.

All enrolled Scoli-RISK-1 participants will be re-consented and asked to return for a 5 year FU visit.

DETAILED DESCRIPTION:
Although the incidence of complications in patients undergoing correction of their spinal deformity has been reported extensively, the majority of these studies were retrospective. There were only five studies, three from a single institution, with prospectively collected data that specifically identified complications. The largest series was from Buchowski et al who reported on 108 patients with fixed sagittal deformity undergoing Pedicle Subtraction Osteotomy (PSO) with a 14% over-all complication rate with motor weakness in 11 patients and neurogenic bladder in one patient, of which 3 were permanent. Yang reported on 35 patients undergoing PSOs with a 46% over-all complication rate and one transient nerve root motor deficit. As in 2002 reported on 83 patients undergoing various osteotomies for sagittal imbalance and reported a 34% over-all complication rate with 3 permanent and 3 transient nerve root deficits.

Given this lack of information, there is a need to determine the true incidence of complications using a prospective multi-center design. There is a need to identify neurologic deficits in a more systematic fashion to include spinal cord, cauda equina and nerve root deficits as well as radiculopathies. The risk factors associated with the occurrence of a complication, especially a neurologic complication, also needs to be more fully elucidated. This is increasingly relevant, as newer surgical techniques allow for more aggressive correction of the spinal deformity that may put the spinal cord and nerve roots at increased risk. Valid data on the incidence and types of neurologic deficits is also needed in order to study newer drugs that are available that may mitigate this risk.

The primary objectives of this study are: (i) to establish the incidence of neurologic deficit in "high risk" adult patients undergoing correction of their spinal deformity of adult spinal deformity and (ii) to identify characteristics associated with increased risk of neurologic complications. Secondary objectives include (i) to determine the incidence of all complications related to surgical correction of "high risk" adult spinal deformity; (ii) to determine the short-term clinical outcomes in patients undergoing correction of their spinal deformity and (iii).to determine amount of radiographic and clinical correction of deformity

ELIGIBILITY:
Inclusion Criteria:

* Participant completed Scoli-RISK-1 study (no withdraws or drop-outs)
* Signed informed consent for extended study

Exclusion Criteria:

* Subjects enrolled in Scoli-RISK-1 which are unlikely to comply with the FU
* Subjects which by law are not eligible to participate any longer in clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant completed Scoli-RISK-1 study are potential subjects for this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Rate of neurologic complication | 5 years postoperative
  Rate of treatment-related neurological complications determined by the Clinical Endpoint Committee (CEC) whether complications are of neurological nature or not.
Absolute change in motor status as measured by the ASIA LEMS | between baseline and 5 years postoperative

SECONDARY OUTCOMES:
ASIA Sensory Score | Change between baseline and 5 years postoperative
  Sensory status as measured by the ASIA Sensory Score
ASIA Impairment Scale | Change between baseline and 5 years postoperative
  Neurological status as measured by the ASIA Impairment Scale
SRS-22R | Change between baseline and 5 years postoperative
  Function, pain and self-image as measured by the SRS-22R
ODI v2.1a | Change between baseline and 5 years postoperative
  Functional impairment as measured by the ODI v2.1a score
SF-36 v2.0 | Change between baseline and 5 years postoperative
  Quality of life as measured by the SF-36 v2.0
Radiographic measures | Change between baseline and 5 years postoperative
  major coronal curve, coronal balance, sagital alignment, T2-T12 sagital cobb, T12-S1 sagital cobb, major sagital curve

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lenke, MD, Principal Investigator — Scoliosis Research Society
Locations (11):
- United States (5):
  - University of California, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - Department of Orthopaedic Surgery, Washington University School of Medicine, St Louis, Missouri
  - NYU School of Medicine, New York, New York
  - University of Virginia, Charlottesville, Virginia
- University of Toronto Hospital, Toronto, Ontario, Canada
- China (2):
  - University of Hong Kong, Hong Kong
  - Nanjing Drum Tower Hospital, Nanjing
- Hamamatsu University School of Medicine, Hamamatsu, Japan
- Hospital Universitari Vall D'Hebron, Barcelona, Spain
- University Hospital Nottingham, NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.aospine.org
- See also: Related Info — http://www.srs.org/